CLINICAL TRIAL: NCT00293488
Title: An Open Label Phase I Study Evaluating Safety, Tolerability and Pharmacokinetics of SL-11047 in Patients With Refractory Lymphoma
Brief Title: SL-11047 in Treating Patients With Relapsed or Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Progen Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: PROGEN-SL002; CDR0000463738 (Registry Identifier: PDQ (Physician Data Query)); UCSF-H1956-21906-02; UCSF-SL002
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
Keywords: anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome | interventions — (N(1),N(12))bis(ethyl)-6,7-dehydrospermine

INTERVENTIONS:
Drug: polyamine analogue PG11047

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as SL-11047, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of SL-11047 in treating patients with relapsed or refractory lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of SL-11047 in patients with relapsed or refractory lymphoma.
* Describe and quantify the toxicity of SL-11047 administered to patients with relapsed or refractory lymphoma.

Secondary

* Describe the pharmacokinetics of SL-11047 administered as a 30-minute IV infusion.
* Assess the response rate and duration of response in patients treated with SL-11047.
* Assess the level of SL-11047 within tumor tissues following intravenous administration of the drug.
* Determine the sensitivity of abnormal circulating macrophages to SL-11047.

OUTLINE: This is an open-label, nonrandomized, dose-escalation study.

Patients receive SL-11047 IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SL-11047 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* confirmed Hodgkin's or non-Hodgkin's lymphoma (NHL) of any histology

  * The following NHL types are eligible:

    * Diffuse large B-cell lymphoma
    * Follicular lymphoma
    * Mantle Cell lymphoma
    * Marginal zone lymphoma (including lymphoma of mucosa-associated tissue [MALT])
    * Anaplastic large cell lymphoma
    * Peripheral T-cell lymphoma
    * Cutaneous T-cell lymphoma
    * T/NK cell lymphoma
    * Angioimmunoblastic lymphadenopathy-type T-cell lymphoma
    * Burkitt's lymphoma NOTE: * If histologic confirmation was made at initial diagnosis, confirmation of relapsed or refractory disease can be made by repeat histologic evaluation OR by evidence of regrowth at a site of disease that was previously histologically confirmed
* Relapsed after or refractory to ≥ 2 prior therapeutic regimens OR patient is ineligible to receive potentially curative therapy
* Bidimensionally measurable or evaluable (e.g., bone marrow or infiltrative organ involvement) disease by physical exam or radiographic study
* No suspicion or evidence of lymphomatous meningitis

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* ECOG performance status 0-4
* Not pregnant
* Negative pregnancy test
* Fertile patients must use medically prescribed contraception
* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count ≥ 50,000/mm^3*
* Hemoglobin ≥ 8 g/dL*
* Serum creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 mg/dL**
* Transaminases < 5 times upper limit of normal**
* No other malignancy within the past 5 years other than curatively treated non-metastatic skin cancer or in situ cervical carcinoma
* No history of significant or symptomatic cardiac arrhythmia
* No history of myocardial infarction
* No significant ventricular conduction abnormality by ECG or Holter monitoring, as evidenced by any of the following:

  * Prior myocardial infarction
  * Three or more premature ventricular contractions in a row
* No history of pancreatitis
* No history of recent gastrointestinal bleeding

  * Must have heme-negative stool at enrollment NOTE: *Cytopenias due to direct lymphomatous involvement allowed

NOTE: **Elevated due to direct lymphomatous involvement allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy
* Recovered from prior chemotherapy (alopecia or anemia allowed)
* More than 3 weeks since prior investigational drugs
* No prophylactic antiemetics during course 1
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hicks — Progen Pharmaceuticals
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States